CLINICAL TRIAL: NCT00808769
Title: Comparison of Prilosec OTC® Versus Zegerid® for Gastric Acid Suppression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 2008122
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Normal Healthy Subject Population
MeSH Terms: interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Zegerid®
  Interventions: Drug: Zegerid®
- 2 (Experimental): Prilosec OTC®
  Interventions: Drug: Prilosec OTC®

INTERVENTIONS:
Drug: Zegerid® — capsule(20 mg omeprazole/sodium bicarbonate), single dose
  Arms: 1
Drug: Prilosec OTC® — Omeprazole-magnesium 20.6 mg, tablet, single dose
  Arms: 2

SUMMARY:
The purpose of this study is to compare Prilosec OTC® and Zegerid® in their effects on gastric acid suppression.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects who are 18-65 years of age;
* Non-childbearing potential females or those using birth control

Exclusion Criteria:

* History of significant GI disease
* Any significant medical illness
* History of hypersensitivity, allergy or intolerance to omeprazole or other proton pump inhibitors;
* Currently using GI medications
* GI disorder or surgery leading to impaired drug absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McRorie, PhD, FACG, AGAF, Study Director — Procter and Gamble
Locations (1):
- Research Site, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period of this study was November 25 to December 21, 2008
Groups:
- Zegerid® Then Prilosec OTC®: Zegerid® (20 mg omeprazole/sodium bicarbonate) then Prilosec OTC® (20.6 mg omeprazole magnesium)
- Prilosec OTC® Then Zegerid®: Prilosec OTC® (omeprazole magnesium 20.6 mg) then Zegerid® (20 mg omeprazole/sodium bicarbonate)
Period: First Intervention
Arm/Group | Zegerid® Then Prilosec OTC® | Prilosec OTC® Then Zegerid®
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Zegerid® Then Prilosec OTC® | Prilosec OTC® Then Zegerid®
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants] — The study was a cross-over study with 30 subjects receiving each treatment; therefore, baseline characteristics are identical for each treatment.
  participants
    United States | 30

OUTCOME MEASURES:

1. Primary Outcome: The Mean Percent Time Gastric pH > 4.0 on Day 1
Description: In this study, there was evidence of gastric pH probe failure and a high incidence of biologically improbable pH measurements (sustained pH < 1.0) that bring the validity of the results into question. The results of this study are, therefore, inconclusive.
Time Frame: continuously over a 24 hour period
Population: Zeros are entered because the data are corrupted for 2 reasons: probe calibration failure rate was ~10x higher than historically documented, and the probes that calibrated had a high incidence of prolonged pH < 1.0 (highly physiologically improbable). This calls into question the credibility and interpretability of all the pH data.
Arm/Group | Zegerid® Then Prilosec OTC® | Prilosec OTC® Then Zegerid®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Zegerid® Then Prilosec OTC® | Prilosec OTC® Then Zegerid®
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Results of this study were uninterpretable as noted in the Analysis Population Description.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other